CLINICAL TRIAL: NCT00113776
Title: A Multicenter, Open-label, Single Arm Clinical Trial to Determine the Safety of ABX-EGF Extended Therapy in Subjects With Metastatic Colorectal Cancer
Brief Title: Evaluating ABX-EGF Extended Therapy in Subjects With MetastaticColorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030194
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Colorectal Cancer
Keywords: Metastatic Colorectal Cancer, Colon; Colorectal, Rectal Cancer, EGFr; Metastatic, Cancer, ABX-EGF; Panitumumab, Clinical Trial; Immunex, Abgenix, Amgen
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Panitumumab

INTERVENTIONS:
Drug: ABX-EGF

SUMMARY:
The purpose of this study is to examine the safety of ABX-EGF administered as monotherapy in subjects with metastatic colorectal cancer who were previously randomized to best supportive care (BSC) in protocol 20020408 and subsequently determined to have progressive disease.

ELIGIBILITY:
Inclusion Criteria: - Subject previously randomized to BSC in protocol 20020408 and subsequently determined to have progressive disease - ECOG performance status of 0, 1 or 2 - Adequate hematologic, renal and hepatic function Exclusion Criteria: - Myocardial infarction in time interval between completing 20020408 and enrollment in study - History or evidence of interstitial pneumonitis or pulmonary fibrosis - Prior anti-tumor therapies including prior experimental agents or approved anti-tumor small molecules and biologics during the time interval between completing 20020408 protocol and enrollment in this study - Use of systemic chemotherapy or radiotherapy during the time interval between completing 20020408 protocol and enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Incidence of Adverse events
Changes in Lab values
Incidence of HAHA formation

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Van Cutsem E, Siena S, Humblet Y, Canon JL, Maurel J, Bajetta E, Neyns B, Kotasek D, Santoro A, Scheithauer W, Spadafora S, Amado RG, Hogan N, Peeters M. An open-label, single-arm study assessing safety and efficacy of panitumumab in patients with metastatic colorectal cancer refractory to standard chemotherapy. Ann Oncol. 2008 Jan;19(1):92-8. doi: 10.1093/annonc/mdm399. Epub 2007 Sep 4. PMID 17785764
- [Derived] Safari M, Esmaeili H, Mahjub H, Roshanaei G. Estimation of treatment effect in presence of noncompliance and competing risks: a simulation study. Sci Rep. 2023 Aug 18;13(1):13477. doi: 10.1038/s41598-023-40538-2. PMID 37596461
- [Derived] Amado RG, Wolf M, Peeters M, Van Cutsem E, Siena S, Freeman DJ, Juan T, Sikorski R, Suggs S, Radinsky R, Patterson SD, Chang DD. Wild-type KRAS is required for panitumumab efficacy in patients with metastatic colorectal cancer. J Clin Oncol. 2008 Apr 1;26(10):1626-34. doi: 10.1200/JCO.2007.14.7116. Epub 2008 Mar 3. PMID 18316791
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20030194.pdf
- See also: FDA-approved Drug Labeling — http://www.vectibix.com/